CLINICAL TRIAL: NCT02917850
Title: Impact of Hip Flexors Isokinetic Strengthening on Gait Capacities in Subacute Stroke Patients
Acronym: ISOKINETIC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: sponsor decision
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015_32; 2016-A00366-45 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-09-22; First posted 2016-09-28 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Stroke; Hemiplegia; Gait
Keywords: stroke; gait; hip flexors; paresis; hemiplegia
MeSH Terms: conditions — Stroke; Hemiplegia; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isokinetic (Active Comparator): Patients who benefit from the hip flexors isokinetic strengthening rehabilitation program
  Interventions: Procedure: Isokinetic hip flexors strengthening; Procedure: Conventional rehabilitation
- Control (Active Comparator): Patients who benefit from a conventional rehabilitation program
  Interventions: Procedure: Conventional rehabilitation

INTERVENTIONS:
Procedure: Isokinetic hip flexors strengthening — Isokinetic excentric strengthening of paretic hip flexors, 3/w during 6 weeks, in addition to conventional rehabilitation 7/w.
  Arms: Isokinetic
Procedure: Conventional rehabilitation — Conventional rehabilitation 10/w during 6 weeks

SUMMARY:
Post-stroke patients often present with gait disorders due to several physical impairments. Hip flexor deficit is one of the more prevalent trouble and is associated with gait capacities. This study aims at evaluating the impact of an isokinetic hip flexors strengthening rehabilitation program in the subacute phase after stroke. Patients will be randomized to an intervention group (isokinetic rehabilitation) or a control group (conventional rehabilitation) and assessed at the end of the rehabilitation program, at 3 and at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from a first ever stroke
* At the subacute phase
* Able to walk at least 10m with or without assistive devices
* Hip flexors strength on the paretic side > 2/5 (MRC)

Exclusion Criteria:

* Uncontrolled epilepsy
* Contraindications to physical activity (severe arterial hypertension, aortic valvulopathy, severe PAD...)
* History of muscular or joint disorders on the paretic hip
* Subject unable to deliver an informed written consent (due to aphasia, cognitive or psychiatric disorders...)
* Protected persons
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Max gait speed (m/s) | 6 weeks
  Gait speed will be assessed in the 10m walk test

SECONDARY OUTCOMES:
Max gait speed (m/s) | 3 and 6 months
  Gait speed will be assessed in the 10m walk test
Hip flexors strength | 6weeks; 3 and 6 months
  Hip flexors strength will be evaluated using an isokinetic dynamometer (concentric, 30°/s) and motor testing (medical research council)
Gait endurance | 6 weeks; 3 and 6 months
  Gait endurance will be assessed using the 6MWT
Gait capacities | 6 weeks; 3 and 6 months
  Functional ambulation categories (FAC)
Balance and postural control | 6 weeks; 3 and 6 months
  Postural Assessment for Stroke Scale (PASS)
Balance and postural control | 6 weeks; 3 and 6 months
  Timed-up and go test
Rate of perceived exhaustion during gait | 6 weeks; 3 and 6 months
  Borg scale

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Allart, MD, Principal Investigator — University Hospital, Lille

IPD SHARING:
Plan to Share IPD: Undecided